CLINICAL TRIAL: NCT02607566
Title: Yoga as a Complementary Therapy for Type 2 Diabetes: An Initial Investigation
Brief Title: Yoga as a Complementary Therapy for Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: University of Massachusetts, Lowell (Other); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT008830 (NIH)
Record Dates: First submitted 2015-11-12; First posted 2015-11-18 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2015-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Yoga; Walking; Stress; exercise; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iyengar Yoga (Experimental): Iyengar Yoga Intervention twice weekly for 60 minutes for 12 weeks.
  Interventions: Behavioral: Yoga
- Standard Exercise Program (Active Comparator): professionally supervised program of aerobic exercise including use of an indoor walking track, treadmills, stationary bicycles and elliptical machines, held for 60 minutes twice weekly for 12 weeks
  Interventions: Behavioral: Standard Exercise Program

INTERVENTIONS:
Behavioral: Yoga
  Arms: Iyengar Yoga
Behavioral: Standard Exercise Program — twice weekly aerobic exercise program, 60 minutes for 12 weeks
  Arms: Standard Exercise Program

SUMMARY:
This study will examine the feasibility and acceptability of a twice weekly yoga program for adults with type 2 diabetes. Changes in perceived stress, salivary cortisol, and HbA1c will also be examined.

DETAILED DESCRIPTION:
The purpose of the current proposal is to test a yoga intervention for adults with T2DM and to gather data on the feasibility and acceptability of yoga compared to a contact control for glycemic control. The investigators will conduct a pilot randomized controlled study with participants randomly assigned to 1) Yoga intervention, or 2) A standard exercise (SE) group program (comparison-control). Focus groups will be conducted with participants at the end of the intervention to identify facilitators and barriers to yoga practice and to examine their perceptions and beliefs about yoga and its relationship to stress and diabetes management. The investigators will explore the effect of yoga on stress (biomarker = salivary cortisol) that may act as a mechanism of action underlying the efficacy of yoga for improved glycemic control. The investigators will also measure HbA1c levels, fasting and postprandial plasma glucose at baseline, end of treatment (12-weeks), 6- and 9-month follow-ups. Study feasibility and acceptability will be assessed using participant recruitment, attendance and retention rates, and compliance with study protocols and satisfaction with the program. Participants will also attend a focus-group discussion of the program at the end of treatment. Results from this study will provide scientific basis for a future larger clinical trial. Yoga, if found to offer advantages for glycemic control, can have potential for high impact on current practices of diabetes management.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for more than 6 months
* HbA1c > 6.5
* Body Mass Index < 42

Exclusion Criteria:

* Serious co-morbid condition (e.g. uncontrolled hypertension, glaucoma, heart failure)
* Complications of diabetes (e.g. diabetic retinopathy, neuropathy, nephropathy)
* Serious psychiatric disorder (e.g. psychosis, major depression, panic attacks, suicidality, or substance dependence)
* Body Mass Index of 42 or greater
* Pregnancy or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Acceptability as measured by session attendance | 12 weeks
  Number of sessions attended
Feasibility as measured by study completion | 6 months
  Percent of enrolled subjects completing all assessments

SECONDARY OUTCOMES:
Changes in diabetes-related distress as measured by Diabetes Related Distress Survey | Baseline to Week 12
  Percent change in score on the Diabetes Related Distress Survey (Polonsky et al., 1995)
Changes in Salivary Cortisol (ug/dL) between baseline and week 12 | Baseline to Week 12
  Saliva samples collected at baseline and week 12 will be assayed for cortisol levels (ug/dL)
HbA1c | 6 months
  HbA1c levels from blood draws
Diabetes Self-Care | 12 weeks
  Surveys of diabetes related self care activities

CONTACTS AND LOCATIONS:
Overall Officials: Beth Bock, PhD, Principal Investigator — The Miriam Hospital
Locations (2):
- United States (2):
  - The Miriam Hospital- CORO building, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Thind H, Fava JL, Guthrie KM, Stroud L, Gopalakrishnan G, Sillice M, Gidron N, Bock BC. Yoga as a Complementary Therapy for Adults with Type 2 Diabetes: Design and Rationale of the Healthy, Active, and in Control (HA1C) Study. Int J Yoga Therap. 2018 Nov;28(1):123-132. doi: 10.17761/2018-00026. Epub 2018 Aug 21. PMID 30130144
- [Result] Thind H, Guthrie KM, Horowitz S, Conrad M, Bock BC. "I can do almost anything": The experience of adults with type 2 diabetes with a yoga intervention. Complement Ther Clin Pract. 2019 Feb;34:116-122. doi: 10.1016/j.ctcp.2018.11.011. Epub 2018 Nov 16. No abstract available. PMID 30712714
- [Result] Bock BC, Thind H, Fava JL, Dunsiger S, Guthrie KM, Stroud L, Gopalakrishnan G, Sillice M, Wu W. Feasibility of yoga as a complementary therapy for patients with type 2 diabetes: The Healthy Active and in Control (HA1C) study. Complement Ther Med. 2019 Feb;42:125-131. doi: 10.1016/j.ctim.2018.09.019. Epub 2018 Sep 26. PMID 30670230
- [Result] Thind H, Lantini R, Balletto BL, Donahue ML, Salmoirago-Blotcher E, Bock BC, Scott-Sheldon LAJ. The effects of yoga among adults with type 2 diabetes: A systematic review and meta-analysis. Prev Med. 2017 Dec;105:116-126. doi: 10.1016/j.ypmed.2017.08.017. Epub 2017 Sep 4. PMID 28882745